CLINICAL TRIAL: NCT03251417
Title: Apatinib and Irinotecan Combination Treatment in Unresectable or Metastatic Esophageal Squamous Cell Carcinoma Patients Failed in First-line Chemotherapy: A Phase II Study
Brief Title: Apatinib and Irinotecan Combination Treatment in Unresectable or Metastatic Esophageal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because PD-1 antibodies had been proved to be a standard second-line treatment in esophageal cancer, the potential benefit of present intervention is under re-evaluation.
Sponsor: Peking University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xiaodong Zhang, Associated Professor of the VIP2 GI Division of Medical Department, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBE002
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Irinotecan; Apatinib
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Irinotecan; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination treatment (Experimental): Combination treatment of irinotecan and apatinib.
  Interventions: Drug: Irinotecan; Drug: Apatinib

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 150mg/m2, repeated very 2 weeks for 3 to 6 cycles.
  Other Names: CPT-11
Drug: Apatinib — Apatinib 500 mg oral take, daily
  Other Names: YN968D1

SUMMARY:
Esophageal cancer is a common malignant disease worldwide especially in china. Though esophagectomy and definitive chemoradiotherapy are standard treatments, disease relapses in many patients and the prognosis of metastatic ESCC is still poor. For patients with unresectable or metastatic ESCC, chemotherapy is an important treatment alone or with radiotherapy. Taxane, platinum, and fluoropyrimidine have been reported effective in ESCC and is used as first-line treatment of ESCC. As for 2nd-line treatment, both irinotecan and taxane had been recommended based on data from clinical trials which were most enrolled esophageal or esophageal-gastric junction adenocarcinoma and with only small sample size. Therefore, it is still urgently needed to explore effective 2nd-line treatment for ESCC.

Apatinib, also known as YN968D1, is an orally antiangiogenic agents. Preclinical and clinical data had shown that it is effective in the treatment of a variety of solid tumors including esophageal cancer. It had been approved as a 3rd-line treatment for patients with advanced gastric cancer by state FDA of China in 2014. And the safety data showed that hemorrhage is rare and non-fetal which is different from bevacizumab.

Therefore, the investigators initialize this phase II study to explore the efficacy and safety of irinotecan and apatinib combination treatment in unresectable or metastatic ESCC patients who failed in 1st-line chemotherapy or chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years. Both genders are eligible.
* Patients must have histologically confirmed esophageal squamous cell carcinoma with unresectable or metastatic disease.
* With measurable or evaluable disease defined by RECIST 1.1 criteria by multi-slice spiral CT or MR scan.
* Failed in or disease progressed after fist-line chemotherapy (A. If failed in preoperative chemotherapy / chemoradiotherapy or disease progressed in 24 weeks after esophagectomy, the preoperative chemotherapy/ chemoradiotherapy is regard as first-line chemotherapy. B. If failed in definitive chemoradiotherapy or disease progressed in 24 weeks after definitive chemoradiotherapy, the definitive chemoradiotherapy is regard as first-line chemotherapy; C. If failed in or relapse in 24 weeks after adjuvant chemotherapy, the adjuvant chemotherapy is regard as first line chemotherapy).
* Patients must have a performance status of 0-2 on the ECOG scale.
* Life expectancy ≥3 months.
* With normal marrow, liver and renal function:a hemoglobin (HGB) of ≥110g/L (without blood transfusion during 14 days); a neutrophil count of ≥2.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL) or ≤3 UNL in case of liver metastasis. a creatinine (Cr) of ≤ 1.5 UNL or a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis. Fecal occult blood (-); Urine test: protein<(++) or <1.0g per 24 hours.
* Without bleeding and thrombosis disease.
* With normal coagulation function: APTT, PT and INR, each ≤ 1.5 ULN
* With normal electrocardiogram results and no history of congestive heart failure.
* Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug.
* With good compliance and agree to accept follow-up of disease progression and adverse events.
* With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.

Exclusion Criteria:

* Patients who have received irinotecan or apatinib in previous treatment.
* Other pathological type cancers of esophagus except for squamous cell carcinoma
* Uncontrolled hypertension (Treatment of antihypertensive drugs cannot reduced to the normal range: systolic pressure ≤140 mmHg and diastolic pressure ≤90 mmHg)
* With ≥grade 2 coronary heart disease, arrhythmia (including QTc interval prolongation male >450 ms, women >470 ms)
* Cannot take oral tables including uncontrolled vomiting, chronic diarrhea and intestinal obstruction.
* With potential bleeding risk of GI including (1) peptic ulcer and fecal occult blood (++ - +++); (2) melena or hematemesis history in last 3 months;(3) In case of fecal occult blood (+) or (+/-),fecal occult blood examination must be repeat in one week. If fecal occult blood is still (+) or (+/-),endoscopy is required and if there are ulcer or other diseases with bleeding risk in the opinion of the investigators. (4) Primary tumour lesion is of deep ulcer and in the opinion of the investigators may place the patient at risk of fetal bleeding or GI perforation.
* Urine test: protein>(++) or >1.0g per 24 hours.
* With abnormal coagulation function (INR>1.5 ULN, APTT>1.5 ULN),
* With thrombosis or receiving anticoagulant treatment.
* With serious diseases such as congestive heart failure, uncontrolled myocardial infarction and arrhythmia, liver failure and renal failure.
* With brain metastasis
* Pregnant or lactated women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Disease control rate | From enrollment to 3 months after treatment.
  The percentage of patients with CR, PR, and SD response after 3 cycles' treatment according to RESIST v1.1 criteria.

SECONDARY OUTCOMES:
Safety: All reported adverse events (NCI CTCAE 4.0 criteria) | From enrollment to progression of disease or 1 months after treatment.
  All reported adverse events (NCI CTCAE 4.0 criteria) during treatment and one months after treatment.
Objective response rate | From enrollment to 3 months after treatment
  Clinical response rate of treatment (CR+PR) according to RESIST v1.1 criteria
Median progression-free survival time | From enrollment to progression of disease. Estimated time is about 4 months
  The length of time from enrollment until the time of progression of disease
Median overall survival time | From enrollment to death of patients, estimated about 8 months.
  The length of time from enrollment until the time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jia, M.D., Principal Investigator — Beijing Cancer Hospital/ Peking University Cancer Hospital
Locations (1):
- Beijing Cancer Hospital / Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided